CLINICAL TRIAL: NCT01574157
Title: Investigations of the Optimum Serum Bicarbonate Level in Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-002-11F
Record Dates: First submitted 2012-03-27; First posted 2012-04-10 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Renal Insufficiency; Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Bicarbonate (Active Comparator): Participants were prescribed 0.5 meq of sodium bicarbonate per 1 kilogram of lean body weight daily for six months
  Interventions: Drug: Sodium bicarbonate
- Placebo (Placebo Comparator): Participants were prescribed an identical number of placebo tablets had they been assigned to the intervention, and took this daily for six months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium bicarbonate — Participants will receive 0.5 meq of sodium bicarbonate per 1 kilogram of lean body weight daily. The total amount will be divided into twice daily doses.
  Arms: Sodium Bicarbonate
Drug: Placebo — Participants will receive an identical number of placebo tablets had they been assigned to the intervention. Placebo will be divided into twice daily doses and receive this for six months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if treatment with sodium bicarbonate will lower urine levels of proteins that are indicators of kidney damage in people with diabetes who also have chronic kidney disease.

DETAILED DESCRIPTION:
Diabetic chronic kidney disease (CKD) is a common problem in Veterans and progresses to end-stage renal disease in many people. It is important to identify treatment strategies that will help prevent the progression of CKD to overt kidney failure. The purpose of this study is to see if sodium bicarbonate reduces urinary markers of kidney damage in Veterans with diabetic CKD and normal serum bicarbonate levels.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age older than 18 years
* Diabetes mellitus
* Serum bicarbonate 22 - 28 mmol/L on the most recent measurement within the past six months
* Stage 2, 3, or 4 CKD (defined as estimated glomerular filtration rate (eGFR) 15 - 89 ml/min/1.73m2 using the CKD-Epidemiology equation)
* Urinary albumin:creatinine ratio > 30 mg/gm on the most recent sample within the past 12 months.

Exclusion Criteria:

* Lean body weight > 100 kg
* Use of oral medications typically prescribed to raise low serum bicarbonate levels (i.e. sodium bicarbonate, sodium citrate, potassium citrate).
* Serum potassium < 3.5 meq/L at enrollment visit
* Use of 5 or more antihypertensive agents, regardless of the indications of each agent
* Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at the enrollment or baseline visit
* Diagnosis of congestive heart failure with current, active Class III or IV New York Heart Association symptoms.
* Significant fluid overload such that it is unsafe in the opinion of the PI for the patient to participate in the trial
* chronic gastrointestinal disorder or any other factors judged to be likely to limit adherence to interventions (i.e. alcoholism, a history of missing clinic visits)
* Chronic immunosuppressive therapy for transplanted organs or other indications
* Individuals who are currently a member of a vulnerable population (I.e. incarcerated, pregnant).

  11.Currently participating in another interventional research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalani L Raphael, MD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gardner J, Tuttle K, Raphael KL. Influence of Medications Containing Acid Salts on Serum Bicarbonate in CKD. Kidney360. 2020 Mar 31;1(5):330-336. doi: 10.34067/KID.0000532019. eCollection 2020 May 28. PMID 35369374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from VA Salt Lake City Healthcare System from November 2012 to October 2017.
Period: Overall Study
Arm/Group | Sodium Bicarbonate | Placebo
Started | 35 | 39
Month 3 | 31 | 33
Completed (Month 6) | 31 | 31
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate | Placebo | Total
Number analyzed (Participants) | 35 | 39 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 73 (8) | 72 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 34 | 38 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 32 | 35 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 32 | 36 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 39 | 74
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m2] | 50 (20) | 52 (16) | 51 (18)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 129 (12) | 127 (11) | 128 (12)
Use of angiotensin converting enzyme-inhibitor (ACE-I) or angiotensin receptor blocker (ARB) [Count of Participants; unit: Participants] | 28 | 34 | 62
Total body weight [Mean (Standard Deviation); unit: kg] | 100 (18) | 101 (22) | 101 (20)
Lean body weight [Mean (Standard Deviation); unit: kg] | 67 (8) | 68 (9) | 68 (9)
Congestive heart failure [Count of Participants; unit: Participants] | 1 | 4 | 5
Serum total carbon dioxide (CO2) [Mean (Standard Deviation); unit: meq/L] | 24 (3) | 24 (2) | 24 (2)
Serum potassium [Mean (Standard Deviation); unit: meq/L] | 4.2 (0.4) | 4.3 (0.4) | 4.2 (0.4)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 7.5 (1.0) | 7.6 (1.3) | 7.5 (1.1)
Urinary albumin/creatinine [Median (Inter-Quartile Range); unit: mg/g] | 121 [84 to 412] | 131 [46 to 324] | 121 [58 to 370]
Urinary pH [Mean (Standard Deviation); unit: units on a scale] | 5.6 (0.4) | 5.4 (0.4) | 5.5 (0.4)
Urinary ammonium [Mean (Standard Deviation); unit: meq/d] | 36 (18) | 33 (21) | 34 (20)
Urinary titratable acids [Mean (Standard Deviation); unit: meq/d] | 32 (14) | 31 (16) | 32 (15)
Urinary transforming growth factor-B1/creatinine [Median (Inter-Quartile Range); unit: ng/g] | 122 [79 to 186] | 103 [68 to 147] | 112 [74 to 157]
Urinary kidney injury molecule-1/creatinine [Median (Inter-Quartile Range); unit: ng/mg] | 0.91 [0.57 to 1.87] | 0.88 [0.59 to 1.89] | 0.89 [0.58 to 1.87]
Urinary fibronectin/creatinine [Median (Inter-Quartile Range); unit: ng/mg] | 107 [75 to 194] | 97 [65 to 147] | 102 [74 to 173]
Urinary neutrophil gelatinase-associated lipocalin/creatinine [Median (Inter-Quartile Range); unit: ng/mg] | 10.5 [7.0 to 23.6] | 11.9 [6.3 to 24.0] | 11.1 [6.5 to 23.8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Transforming Growth Factor Beta 1 (TGF-b1)
Description: Urinary TGF-b1 is considered a marker of renal fibrosis
Time Frame: The mean of the 3-month and 6-month urinary TGF-b1 measurement will be compared to the baseline value between the groups.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 35 | 39
percent change | 7.6 [-9.6 to 28.0] | -4.4 [-19.4 to 13.4]
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Placebo; The primary analysis compared the mean change from baseline in the sodium bicarbonate group to the mean change from baseline in the placebo group; Test type: Superiority; Mean Difference (Final Values) = 12.6, 95% CI 2-sided [-9.6 to 40.1]

2. Secondary Outcome: Change in Urinary Levels of Kidney Injury Molecule-1 (KIM-1)
Description: KIM-1 is a marker of of kidney injury.
Time Frame: The mean of the 3-month and 6-month measurements will be compared to the baseline values between the groups.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 35 | 39
percent change | -11.4 [-33.0 to 17.0] | -1.5 [-24.9 to 29.2]
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Placebo; The main analytic strategy for this secondary outcome was a comparison of the mean change from baseline in the sodium bicarbonate group to the mean change from baseline in the placebo group; Test type: Superiority; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-38.2 to 30.8]

3. Secondary Outcome: Change in Urinary Levels of Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: NGAL is a marker of kidney injury
Time Frame: The mean of the 3-month and 6-month measurements will be compared to the baseline values between the groups.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 35 | 39
percent change | -28.5 [-48.7 to -0.3] | 5.9 [-23.9 to 47.6]
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -32.5, 95% CI 2-sided [-56.3 to 4.2]

4. Secondary Outcome: Change in Urinary Levels of Fibronectin
Description: Fibronectin is a marker of kidney injury.
Time Frame: The mean of the 3-month and 6-month measurements will be compared to the baseline values between the groups.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 35 | 39
percent change | 8.8 [-9.4 to 30.7] | 1.1 [-15.8 to 21.3]
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 7.7, 95% CI 2-sided [-15.1 to 36.5]

5. Secondary Outcome: Change in Urinary Albumin Levels
Description: Urinary albumin is a marker of kidney damage
Time Frame: The mean of the 3-month and 6-month measurements will be compared to the baseline values between the groups.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 35 | 39
percent change | 21.1 [-3.1 to 51.3] | 11.9 [-10.5 to 39.8]
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-24.6 to 35.9]

6. Secondary Outcome: Change in Estimated Glomerular Filtration (eGFR)
Description: eGFR is a measure of kidney function
Time Frame: The mean of the 3-month and 6-month measurements will be compared to the baseline values between the groups.
Measure: Mean (95% Confidence Interval); unit: ml/min per 1.73m2
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 35 | 39
ml/min per 1.73m2 | 1.96 [-0.47 to 4.40] | -1.41 [-3.80 to 0.99]
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 3.37, 95% CI 2-sided [-0.05 to 6.79]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during each participant's 6-month follow-up period.
Arm/Group | Sodium Bicarbonate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/39
Other Adverse Events (participants affected / at risk) | 0/35 | 0/39

LIMITATIONS AND CAVEATS:
Change in urinary levels of Bb and membrane attack complex (MAC) were initial secondary outcomes. However, we had difficulty measuring these. Many subjects could not complete the physical activity assessment, which was an initial secondary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT01574157/Prot_SAP_000.pdf